CLINICAL TRIAL: NCT07395362
Title: A Prospective Single-Arm Study Evaluating the Safety, Feasibility, and Perioperative Recovery of Robot-Assisted Percutaneous Ablation/Localization Combined With Non-Intubated Video-Assisted Thoracoscopic Surgery for Multiple Pulmonary Nodules
Brief Title: Hybrid Robot-Assisted Percutaneous Ablation and Non-Intubated VATS for Multiple Pulmonary Nodules
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, Department of Thoracic Surgery, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GZMUFAH-MLN-HYBRID-2026-01
Record Dates: First submitted 2026-01-25; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-01

CONDITIONS: Multiple Pulmonary Nodules
Keywords: Multiple pulmonary nodules; Ground-glass nodules; Robot-assisted percutaneous ablation; CT-guided intervention; Non-intubated video-assisted thoracoscopic surgery NiVATS
MeSH Terms: conditions — Multiple Pulmonary Nodules

STUDY DESIGN:
Intervention Model Description: This is a prospective, single-arm study in which all enrolled participants receive a predefined hybrid treatment strategy combining robot-assisted percutaneous intervention and non-intubated video-assisted thoracoscopic surgery during the same hospitalization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hybrid Robot-Assisted Percutaneous Intervention Plus Non-Intubated VATS (Experimental): Participants in this single-arm study receive a predefined hybrid treatment strategy during the same hospitalization. The intervention consists of robot-assisted CT-guided percutaneous procedures (including localization, biopsy, and/or thermal ablation as clinically appropriate) for selected pulmonary nodules, followed by non-intubated video-assisted thoracoscopic surgery for resection of the dominant pulmonary lesion. Conversion to conventional intubated anesthesia is permitted if clinically indicated.
  Interventions: Procedure: Hybrid Robot-Assisted Percutaneous Intervention and Non-Intubated Video-Assisted Thoracoscopic Surgery

INTERVENTIONS:
Procedure: Hybrid Robot-Assisted Percutaneous Intervention and Non-Intubated Video-Assisted Thoracoscopic Surgery — This intervention consists of a predefined hybrid procedural strategy performed during the same hospitalization. Selected pulmonary nodules are managed using robot-assisted CT-guided percutaneous procedures, including localization, biopsy, and/or thermal ablation as clinically appropriate. Subsequently, the dominant pulmonary lesion is resected using non-intubated video-assisted thoracoscopic surgery under spontaneous ventilation anesthesia. Conversion to conventional intubated anesthesia is permitted if clinically indicated.
  Other Names: Robot-assisted percutaneous ablation; CT-guided percutaneous localization; Non-intubated VATS; NiVATS

SUMMARY:
The goal of this clinical trial is to evaluate the safety and feasibility of a predefined hybrid treatment strategy in patients with multiple pulmonary nodules who require surgical management of at least one dominant lesion. The strategy combines robot-assisted CT-guided percutaneous ablation and/or localization with non-intubated video-assisted thoracoscopic surgery (NiVATS) performed during the same hospitalization.

The main questions this study aims to answer are:

Is the hybrid treatment strategy associated with an acceptable rate of perioperative serious complications?

Can the planned combination of robot-assisted percutaneous intervention and NiVATS be completed successfully in a real-world clinical setting?

Participants will:

Undergo preoperative evaluation and multidisciplinary assessment;

Receive robot-assisted CT-guided percutaneous ablation and/or localization for selected pulmonary nodules;

Undergo non-intubated video-assisted thoracoscopic surgery for resection of the dominant pulmonary lesion;

Be followed for perioperative outcomes and short-term recovery up to 30 days after surgery.

DETAILED DESCRIPTION:
This is a prospective, single-arm interventional study conducted at a tertiary academic medical center. The study enrolls adult patients with multiple pulmonary nodules, including at least one dominant lesion that meets standard indications for thoracoscopic surgical resection and one or more additional nodules for which complete surgical resection is considered undesirable due to concerns regarding lung parenchymal preservation or procedural risk.

All participants receive a predefined hybrid treatment strategy during the same hospitalization. Selected secondary pulmonary nodules are managed using robot-assisted CT-guided percutaneous procedures, including localization, biopsy, and/or thermal ablation as clinically appropriate. Subsequently, the dominant lesion is resected using non-intubated video-assisted thoracoscopic surgery under spontaneous ventilation anesthesia. Conversion to conventional intubated anesthesia is permitted if clinically indicated.

The primary focus of this study is to assess perioperative safety and technical feasibility rather than comparative efficacy. Safety is evaluated by monitoring perioperative complications within 30 days after the procedure, while feasibility is assessed based on successful completion of the planned hybrid treatment strategy. Secondary observations include perioperative recovery parameters such as length of hospital stay, postoperative pain, and short-term clinical outcomes.

This study is designed to provide prospective evidence regarding the clinical applicability of a hybrid, lung parenchyma-preserving approach for the management of multiple pulmonary nodules within the framework of current surgical and interventional practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 to 85 years at the time of enrollment.
2. Presence of multiple pulmonary nodules identified on chest computed tomography (CT).
3. At least one dominant pulmonary lesion meeting standard indications for thoracoscopic surgical resection based on radiologic assessment.
4. At least one additional pulmonary nodule for which complete surgical resection is considered undesirable due to lung parenchyma preservation concerns or procedural risk, and deemed suitable for robot-assisted CT-guided percutaneous intervention.
5. Determined by a multidisciplinary team (MDT) to be an appropriate candidate for the predefined hybrid treatment strategy.
6. Eligible for non-intubated video-assisted thoracoscopic surgery based on preoperative anesthetic evaluation (ASA physical status I-III).
7. Ability to understand the study procedures and provide written informed consent.

Exclusion Criteria:

1. Pulmonary nodules located centrally or adjacent to major airways, major vessels, or the heart, where safe percutaneous intervention is not feasible.
2. Pure ground-glass nodules with a maximum diameter < 6 mm, for which active surveillance is recommended.
3. Clinical evidence of N1/N2 lymph node involvement or distant metastasis.
4. Severe cardiopulmonary disease, interstitial lung disease, or other conditions that preclude thoracoscopic surgery or anesthesia.
5. Coagulation disorders or ongoing anticoagulation therapy that cannot be safely discontinued.
6. Pregnancy or breastfeeding.
7. Any condition that, in the opinion of the investigator, would make participation unsafe or interfere with study assessments.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2026-08-28 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Perioperative Serious Complications | Within 30 days after the procedure
  The proportion of participants who experience serious perioperative complications within 30 days after the procedure, defined as complications of Clavien-Dindo grade III or higher, including events requiring surgical, endoscopic, or radiologic intervention, intensive care management, or resulting in death.

SECONDARY OUTCOMES:
Successful completion rate of the planned hybrid treatment strategy | From the start of the percutaneous intervention to completion of the planned hybrid procedure during the same hospitalization, assessed up to 30 days
  Technical feasibility is defined as the proportion of participants in whom the planned hybrid treatment strategy-robot-assisted CT-guided percutaneous intervention followed by non-intubated video-assisted thoracoscopic surgery-is successfully completed without unplanned abandonment of the procedure. Conversion to conventional intubated anesthesia is permitted and will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of GZMU, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results reported in publications, including baseline characteristics, perioperative variables, and outcome measures, will be shared. No direct identifiers will be included. Data not relevant to the primary and secondary outcomes will not be shared.
Supporting Information: Study Protocol
Time Frame: The IPD will be available beginning 6 months after publication of the primary study results and will be available for up to 3 years thereafter.
Access Criteria: Access to the de-identified IPD will be granted to qualified researchers who provide a methodologically sound research proposal. Requests should be submitted to the principal investigator and will be reviewed by the study team. Approved researchers will be required to sign a data use agreement before access is granted. Data will be shared through secure data transfer methods.

REFERENCES:
- [Result] Ye X, Fan W, Wang Z, Wang J, Wang H, Niu L, Fang Y, Gu S, Liu L, Liu B, Zhuang Y, Wei Z, Li X, Li X, Li Y, Li C, Yang X, Yang W, Yang P, Lin Z, Meng Z, Hu K, Liu C, Huang Y, Huang G, Huang K, Peng Z, Han Y, Jin Y, Lei G, Zhai B, Li H, Pan J, Filippiadis D, Kelekis A, Pua U, Futacsi B, Yumchinserchin N, Iezzi R, Tang A, Roy SH. Clinical practice guidelines on image-guided thermal ablation of primary and metastatic lung tumors (2022 edition). J Cancer Res Ther. 2022 Sep;18(5):1213-1230. doi: 10.4103/jcrt.jcrt_880_22. PMID 36204866
- [Result] Chen H, Kim AW, Hsin M, Shrager JB, Prosper AE, Wahidi MM, Wigle DA, Wu CC, Huang J, Yasufuku K, Henschke CI, Suzuki K, Tailor TD, Jones DR, Yanagawa J. The 2023 American Association for Thoracic Surgery (AATS) Expert Consensus Document: Management of subsolid lung nodules. J Thorac Cardiovasc Surg. 2024 Sep;168(3):631-647.e11. doi: 10.1016/j.jtcvs.2024.02.026. Epub 2024 Jun 14. PMID 38878052
- [Result] MacMahon H, Naidich DP, Goo JM, Lee KS, Leung ANC, Mayo JR, Mehta AC, Ohno Y, Powell CA, Prokop M, Rubin GD, Schaefer-Prokop CM, Travis WD, Van Schil PE, Bankier AA. Guidelines for Management of Incidental Pulmonary Nodules Detected on CT Images: From the Fleischner Society 2017. Radiology. 2017 Jul;284(1):228-243. doi: 10.1148/radiol.2017161659. Epub 2017 Feb 23. PMID 28240562